CLINICAL TRIAL: NCT00614432
Title: Blood Loss at the Time of First Trimester Surgical Abortion in Anticoagulated Women
Status: Completed | Type: Observational
Sponsor: University of Hawaii (Other)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Bliss Kaneshiro, Associate Professor, University of Hawaii
Other Study IDs: OHSU FAMPLAN 3861
Record Dates: First submitted 2008-01-31; First posted 2008-02-13 (Estimated); Results first posted 2018-12-14 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Blood Loss
Keywords: anticoagulation; surgical abortion
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Women who are anticoagulated.
- 2: Matched case controls.

SUMMARY:
The primary objective of this study is to compare blood loss resulting from surgical termination of pregnancy up to 12 weeks gestation between women who are anticoagulated to therapeutic levels and those who are not anticoagulated. This study is based on the hypothesis that anticoagulant therapy does not increase intraoperative blood loss in women receiving surgical abortions up to 12 weeks gestation.

DETAILED DESCRIPTION:
We intend to conduct a prospective cohort study at Oregon Health and Science University and the University of Hawaii. This study will not be blinded and subjects will not be randomized. Women will be approached about this study after they have made a decision to terminate the pregnancy and have completed the preoperative history and physical examination and surgical consenting process. For patients who are receiving anticoagulant medications, the decision to continue anticoagulant therapy or interrupt it will be made by the patient's physician, independently of this study.

We will recruit women who continue on anticoagulant therapy (heparin, low molecular weight heparin, or warfarin) without interruption for the surgical procedure. Our control group will consist of women who are not on anticoagulant treatment. This is a matched study and our control group will be matched for gestational age, parity, and cesarean section history.

ELIGIBILITY:
Inclusion Criteria:

* Female seeking abortion services
* Less than or equal to 12 weeks gestation
* Age 18-50
* Willing and able to sign informed consent
* Use of Coumadin or LMW heparin (treatment group only)

Exclusion Criteria:

* Unwilling or unable to sign informed consent
* Women taking daily aspirin or herbal therapies containing gingko biloba
* Women with a known history of a bleeding disorder such as von willebrand's disease

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women will be approached about this study after they have made a decision to terminate the pregnancy and have completed the preoperative history and physical examination and surgical consenting process. We will recruit women who continue on anticoagulant therapy (heparin, low molecular weight heparin, or warfarin) without interruption for the surgical procedure. Our control group will consist of women who are not on anticoagulant treatment.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2008-01; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bliss Kaneshiro, M.D., Principal Investigator — University of Hawaii; Alison Edelman, M.D., M.P.H., Principal Investigator — Oregon Health and Science University
Locations (2):
- United States (2):
  - University of Hawaii, Honolulu, Hawaii
  - Oregon Health and Science University, Portland, Oregon

RESULTS

PARTICIPANT FLOW:
Groups:
- Women Who Are Anticoagulated: Women who are anticoagulated having surgical abortion below 12 weeks gestation
- Women Who Are Not Anticoagulated: Women who are not anticoagulated having surgical abortion less than 12 weeks gestation
Period: Overall Study
Arm/Group | Women Who Are Anticoagulated | Women Who Are Not Anticoagulated
Started | 4 | 6
Completed | 4 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Women Who Are Anticoagulated: Women who are anticoagulated.
- Matched Case Controls: Matched case controls.
- Total: Total of all reporting groups
Arm/Group | Women Who Are Anticoagulated | Matched Case Controls | Total
Number analyzed (Participants) | 4 | 6 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 6 | 10
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.0 (7.9) | 23.2 (3.0) | 25.1 (5.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 10
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 6 | 10

OUTCOME MEASURES:

1. Primary Outcome: Volume of Intraoperative Blood Loss
Description: Quantitative blood loss using volume measurement and weight
Time Frame: Post procedure
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | Women Who Are Anticoagulated | Matched Case Controls
Number analyzed (Participants) | 4 | 6
milliliters | 91.5 (88.0) | 52.2 (48.0)

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Women Who Are Anticoagulated | Matched Case Controls
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/6
Other Adverse Events (participants affected / at risk) | 1/4 | 0/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Women Who Are Anticoagulated (N=4) | Matched Case Controls (N=6)
reaspiration (Surgical and medical procedures) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No